CLINICAL TRIAL: NCT04629443
Title: Phase I/II, International, Multicentre, Open-label, Non-randomised, Non-comparative, Study Evaluating the Safety, Tolerability and Clinical Activity of Intravenously Administered S64315, a Selective Mcl-1 Inhibitor, in Combination With Azacitidine in Patients With Acute Myeloid Leukaemia (AML)
Brief Title: Phase I/II Trial of S64315 Plus Azacitidine in Acute Myeloid Leukaemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-64315-004; 2019-004896-38 (EudraCT Number)
Record Dates: First submitted 2020-11-03; First posted 2020-11-16 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukaemia
Keywords: Acute Myeloid Leukaemia; Oncology; Mcl-1 inhibitor; Azacitidine; Combination; Phase I/II; International; Safety; Maximum tolerated dose
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- S64315 (also referred as MIK665) with azacitidine (Experimental)
  Interventions: Drug: S 64315 (also referred as MIK665) and azacitidine

INTERVENTIONS:
Drug: S 64315 (also referred as MIK665) and azacitidine — The combination treatment at the planned doses may be preceded by a 2-week Lead-In Dose period of S64315 (fixed dose) administered via intravenous (IV) infusion over at least 2 hours.
  During the combination treatment period S64315 will be administered according to a dose escalation scheme starting at 50 mg up to 250 mg might be explored. The schedule will be a 21-day cycle with a weekly regimen for S64315 and a daily regimen of azacitidine administered at 75 mg/m² via subcutaneous (SC) injection for 7 days from D1 to D7 of each cycle followed by a rest period of 21 days.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and clinical activity of the combination S64315 with azacitidine in patients with acute myeloid leukaemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years
2. Patients with cytologically confirmed and documented de novo, secondary or therapy-related AML as defined by World Health Organization 2016 classification (Arber, 2016) excluding acute promyelocytic leukaemia (APL, French American-British M3 classification) with: relapsed or refractory disease and without established alternative therapy, or secondary to MyeloDysplastic Syndrome and without established alternative therapy or, newly diagnosed AML, not previously treated for AML and who are not candidate for intensive chemotherapy due to age or comorbidities.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
4. Adequate haematological, renal and hepatic functions based on the last assessment performed within 7 days prior to the first Investigational Medicinal Product administration.

Exclusion Criteria:

1. Previous myeloproliferative syndrome (MPS).
2. Patients previously treated with any Mcl-1 inhibitor.
3. Patients who have not recovered from toxicity of previous anticancer therapy, including Grade ≥ 2 toxicity (except alopecia of any grade) according to the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI CTCAE) version 5.0, prior to the first IMP administration.
4. Severe or uncontrolled active acute or chronic infection.
5. Uncontrolled hepatitis B or C infection.
6. Known carriers of HIV antibodies, history of significant liver disease, active acute or chronic pancreatitis, active central nervous system disease.
7. Troponin > ULN (Upper Limit of reference range) or Troponin T > ULN if Troponin I cannot be assessed.
8. Clinically significant cardiac dysfunction (including New York Heart Association class ≥II heart failure, Left Ventricular Ejection Fraction (LVEF) < 50% as assessed by echocardiography (ECHO) or Multi-Gated Acquisition (MUGA) scan).
9. QT prolongation defined as QTc (QT interval corrected for heart rate) interval (corrected with Fridericia's formula) > 450 ms for males and > 470 ms for females, obtained from triplicate 12-lead ECG.
10. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age.
11. Uncontrolled arterial hypertension (systolic blood pressure (SBP) > 150 mmHg or diastolic blood pressure (DBP) > 95 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- University of Texas MD Anderson Cancer Center Department of Leukemia, Division of Cancer Medicine, Houston, Texas, United States
- Australia (2):
  - Victorian Comprehensive Cancer Centre, Melbourne
  - The Alfred Hospital Malignant Haematology & Stem Cell Transplantation Services, Melbourne
- France (2):
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Saint Antoine, Paris
- Spain (2):
  - H. Universitario Valle de Hebrón Servicio de Hematología, Barcelona
  - H. Universitario La Fe Servicio de Hematologia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH).
  The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg S64315 (Also Referred as MIK665) With Azacitidine; 100 mg S64315 (Also Referred as MIK665) With Azacitidine; 190 mg S64315 (Also Referred as MIK665) With Azacitidine: S 64315 (also referred as MIK665) and azacitidine: The combination treatment at the planned doses may be preceded by a 2-week Lead-In Dose period of S64315 (fixed dose) administered via intravenous (IV) infusion over at least 2 hours.
  During the combination treatment period S64315 will be administered according to a dose escalation scheme starting at 50 mg up to 250 mg might be explored. The schedule will be a 21-day cycle with a weekly regimen for S64315 and a daily regimen of azacitidine administered at 75 mg/m² via subcutaneous (SC) injection for 7 days from D1 to D7 of each cycle followed by a rest period of 21 days.
Period: Overall Study
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Started | 5 | 7 | 5
Completed | 0 | 0 | 0
Not Completed | 5 | 7 | 5
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Progressive Disease | 2 | 3 | 3
Not completed — Physician Decision | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine | Total
Number analyzed (Participants) | 5 | 7 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (8.3) | 60.1 (14.1) | 64.8 (12.9) | 64.9 (12.5)
Age, Customized [Count of Participants; unit: Participants]
  18 to less then 65 | 1 | 4 | 2 | 7
  65 to less then 85 | 4 | 3 | 3 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 7
  Male | 4 | 4 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 7 | 5 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 6 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) (Phase I - Dose Escalation)
Description: Incidence of DLTs starting from the Lead-In Dose period to the end of the first cycle of treatment of S64315 in combination with azacitidine.
Time Frame: Day -13 to Cycle 1 Day 28 (each cycle is 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 3 | 6 | 4
Participants | 0 | 1 | 1

2. Primary Outcome: Number of Adverse Events (AEs) and Severe AEs (Phase I - Dose Escalation)
Description: Incidence and severity of AEs according to NCI CTCAE v5.0
Time Frame: an average of 6 months
Measure: Number; unit: Events
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 5 | 7 | 5
Events
  Total Number of AEs | 72 | 56 | 41
  Number of Severe AEs | 39 | 22 | 13

3. Primary Outcome: Number of Serious Adverse Event (SAEs) and Fatal SAEs (Phase I - Dose Escalation)
Description: Incidence and severity of SAEs according to NCI CTCAE v5.0
Time Frame: Day -13 up to 30 calendar days after the patient's last study visit (an average of 6 months)
Measure: Number; unit: Events
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 5 | 7 | 5
Events
  Total Number of SAEs | 16 | 14 | 5
  Fatal SAEs | 2 | 2 | 0

4. Primary Outcome: Number of Participants With Dose Interruptions (Phase I - Dose Escalation)
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 5 | 7 | 5
Participants
  Dose delay | 3 | 2 | 1
  Dose interruption | 4 | 4 | 3

5. Primary Outcome: Number of Participants With Dose Reductions (Phase I - Dose Escalation)
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 5 | 7 | 5
Participants | 1 | 0 | 0

6. Primary Outcome: Dose Intensity for S64315 (Phase I - Dose Escalation)
Time Frame: Through study completion, an average of 6 months
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 5 | 7 | 5
mg/week | 41.0 (2.7) | 60.3 (19.8) | 119.6 (19.9)

7. Secondary Outcome: Assess Anti-leukemic Activity of S64315 in Combination With Azacitidine (Phase I - Dose Escalation)
Description: Overall survival (OS)
Time Frame: Through study completion, an average of 6 months
Population: In the context of the premature study discontinuation due to strategic reasons, no statistical analyses for this outcome measure was completed since data was not collected.
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Assess Anti-leukemic Activity of S64315 in Combinaison With Azacitidine (Phase I - Dose Escalation)
Description: Duration of response (DOR)
Time Frame: Through study completion, an average of 6 months
Population: as for outcome 7
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Assess Anti-leukemic Activity of S64315 in Combinaison With Azacitidine (Phase I - Dose Escalation)
Description: Best overall response (BOR)
Time Frame: Through study completion, an average of 6 months
Population: as for outcome 7
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Assess Anti-leukemic Activity of S64315 in Combinaison With Azacitidine (Phase I - Dose Escalation)
Description: Progression-free survival (PFS)
Time Frame: Through study completion, an average of 6 months
Population: as for outcome 7
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Assess Anti-leukemic Activity of S64315 in Combinaison With Azacitidine (Phase I - Dose Escalation)
Description: Disease-free survival (DFS)
Time Frame: Through study completion, an average of 6 months
Population: as for outcome 7
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Pharmacokinetic Profile of S64315 Administered in Combination With Azacitidine in Plasma: Area Under the Curve (AUC) (Phase I - Dose Escalation)
Time Frame: At Cycle 1 Day 2 and Cycle 1 Day 9 (each cycle is 28 days)
Population: For Cycle 1 Day 9 in the 50 mg S64315 arm, the blood sample was collected from the same site of IV infusion and therefore, no descriptive statistics were derived due to unreliable PK Data. The other cohorts had less patients analyzed due to missing patient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 3 | 4 | 3
ng.h/mL
  Cycle 1 Day 2 | 1588 (2.9) | 1929 (71) | 7393 (38)
  Cycle 1 Day 9: number analyzed (Participants) | 0 | 1 | 1
  Cycle 1 Day 9 |  | 2235 (NA) — It is not applicable since there was only 1 participant analyzed. | 8584 (NA) — It is not applicable since there was only 1 participant analyzed.

13. Secondary Outcome: Pharmacokinetic Profile of S64315 Administered in Combination With Azacitidine in Plasma: Maximum Concentration (Cmax) (Phase I - Dose Escalation)
Time Frame: At Cycle 1 Day 2 and Cycle 1 Day 9 (each cycle is 28 days)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 3 | 4 | 3
ng/mL
  Cycle 1 Day 2 | 923 (16) | 1021 (59) | 3646 (36)
  Cycle 1 Day 9: number analyzed (Participants) | 0 | 1 | 1
  Cycle 1 Day 9 |  | 1850 (NA) — It is not applicable since there was only 1 participant analyzed. | 4520 (NA) — It is not applicable since there was only 1 participant analyzed.

14. Primary Outcome: Dose Intensity for Azacitidine (Phase I - Dose Escalation)
Time Frame: Through study completion, an average of 6 months
Population: One participant in the 100 mg arm did not receive azacitidine and therefore was not eligible for analysis.
Measure: Mean (Standard Deviation); unit: mg/m^2/week
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
Number analyzed (Participants) | 5 | 6 | 5
mg/m^2/week | 23.5 (17.0) | 18.8 (0.3) | 22.9 (9.1)

ADVERSE EVENTS:
Time Frame: Up to 30 days after the patients last study visit (an average of 6 months)
Arm/Group | 50 mg S64315 (Also Referred as MIK665) With Azacitidine | 100 mg S64315 (Also Referred as MIK665) With Azacitidine | 190 mg S64315 (Also Referred as MIK665) With Azacitidine
All-Cause Mortality (participants affected / at risk) | 2/5 | 5/7 | 2/5
Serious Adverse Events (participants affected / at risk) | 5/5 | 7/7 | 4/5
Other Adverse Events (participants affected / at risk) | 5/5 | 6/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg S64315 (Also Referred as MIK665) With Azacitidine (N=5) | 100 mg S64315 (Also Referred as MIK665) With Azacitidine (N=7) | 190 mg S64315 (Also Referred as MIK665) With Azacitidine (N=5)
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Anorectal cellulitis (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0
Sinusitis aspergillus (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Troponin I increased (Investigations) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg S64315 (Also Referred as MIK665) With Azacitidine (N=5) | 100 mg S64315 (Also Referred as MIK665) With Azacitidine (N=7) | 190 mg S64315 (Also Referred as MIK665) With Azacitidine (N=5)
Alanine aminotransferase increased (Investigations) | 4 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 2
Troponin T increased (Investigations) | 1 | 2 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Administration site erythema (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1
Injection site rash (General disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04629443/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT04629443/SAP_001.pdf